CLINICAL TRIAL: NCT07292779
Title: A Prospective, Clinical Investigation to Evaluate the Performance and Safety of DMFI150 for the Treatment of Nasolabial Folds
Brief Title: A Prospective Clinical Investigation of DMFI150 for Treating Nasolabial Folds
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samyang Biopharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LF15_NLF_EU
Record Dates: First submitted 2025-11-19; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Nasolabial Folds, Wrinkles

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DMFI150 (Experimental): Single injection of DMFI150
  Interventions: Device: DMFI150

INTERVENTIONS:
Device: DMFI150 — Injection of DMFI150 for nasolabial folds.

SUMMARY:
This is a prospective clinical investigation designed to evaluate the performance and safety of DMFI150 for the treatment of nasolabial folds. 30 adult participants will receive a single treatment with the investigational device. The study will assess wrinkle severity using validated aesthetic evaluation scales, as well as overall safety.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18-70 years.
* Score of 3 to 4 on the WSRS (1 = absent, 2 = mild, 3 = moderate, 4 = severe, and 5 = extreme) for both nasolabial folds.
* Able and willing to provide written informed consent.
* Willing to refrain from facial cosmetic procedures during the study.

Exclusion Criteria:

* Use of antiplatelet agents, vitamin E, or NSAIDs within 2 weeks before screening or 2 weeks after treatment.
* History or current bleeding disorders.
* Participation in another clinical trial within 1 month before screening.
* Pregnant or breastfeeding women, or planning pregnancy.
* Women of childbearing potential not using effective contraception.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Wrinkle Severity Rating Scale (WSRS) as Assessed by the Evaluator Investigator (EI) | Baseline to Month 12
  WSRS is a validated 5-point ordinal scale used to evaluate wrinkle severity
  (1 = Absent, 2 = Mild, 3 = Moderate, 4 = Severe, 5 = Extreme). Higher scores indicate more severe wrinkles. The EI will assess the change from baseline to Month 12.

SECONDARY OUTCOMES:
Change from Baseline in Wrinkle Severity Rating Scale (WSRS) Assessed by the Evaluator Investigator (EI) and the Treating Investigator (TI) | Baseline to Month 1,3,6,9,12
  WSRS is a validated 5-point ordinal scale used to evaluate wrinkle severity (1 = Absent, 2 = Mild, 3 = Moderate, 4 = Severe, 5 = Extreme). Higher scores indicate more severe wrinkles. Changes from baseline will be assessed by both EI and TI.
Change from Baseline in Global Aesthetic Improvement Scale (GAIS) Assessed by the Treating Investigator (TI) and by the Subject | Baseline to Month 1,3,6,9,12
  GAIS is a 5-point global improvement scale (3 = Very Much Improved, 2 = Much Improved, 1 = Improved, 0 = No Change, -1 = Worse). Higher scores indicate greater improvement. Both the subject and TI will rate GAIS.
Incidence of Treatment-Related Adverse Events (TRAEs), Adverse Events (AEs), Serious Adverse Events (SAEs), and Device Deficiencies (DDs) | Baseline through Month 12
  All TRAEs, AEs, SAEs, and DDs will be recorded and assessed according to the clinical investigation plan.

CONTACTS AND LOCATIONS:
Locations (1):
- Ocean Clinic, Marbella, Spain

IPD SHARING:
Plan to Share IPD: No